CLINICAL TRIAL: NCT04415450
Title: Effect of Nutrition Education by Health Professionals on Pregnancy Specific Nutrition Knowledge and Healthy Dietary Practice Among Pregnant Women in Asmara, Eritrea
Brief Title: Effect of Nutrition Education on Knowledge and Healthy Dietary Practice Among Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orotta College of Medicine and Health Sciences (Other)
Responsible Party: Principal Investigator, Lidia Ghirmai, Lecturer, Orotta College of Medicine and Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OCMHS
Record Dates: First submitted 2020-05-23; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Pregnancy Nutritional Disease
Keywords: Nutrition education; Knowledge; Practice

STUDY DESIGN:
Intervention Model Description: Pregnant women who were on their first and second trimester of pregnancy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutrition Education Group (Experimental): The experimental group is the group who received the intervention which is the nutrition education and counseling. Phase I of the data collection from the experimental group which is the pregnant women (baseline assessment) using a questionnaire immediately before receiving nutrition counseling from their ANC providers first took place. Health professionals then started providing nutrition education to pregnant women preselected and assessed before the intervention. Immediate post education evaluation of the pregnant women was done by the same questionnaire used to assess in the pretest. Phase II or post intervention data collection of pregnant women was done after the client was appointed for 6 weeks after the counseling session.
  Interventions: Behavioral: Nutrition Education counseling

INTERVENTIONS:
Behavioral: Nutrition Education counseling — In the context of health education program, an educational intervention was developed by the research team based on a training module. The nutrition education contained introductory messages and focused on meanings of healthy diet, eating a variety of food, eating well with the locally available food, hazards of maternal malnutrition, important supplements to be taken during pregnancy, harmful substances to be avoided, and measures of alleviating common discomforts associated with nutrition during pregnancy. The training program was carried out in the form of counseling using printed materials and flip charts for pictorial representation. Self-reading of leaflets containing the core messages for every topic prepared in the native language of the participants was also employed as the women in the study had one each.

SUMMARY:
Healthy pregnancy and birth outcomes is greatly influenced by the intake of adequate and balanced nutrition. Pregnant women's nutritional knowledge and practice have been identified as an important prerequisites for their proper nutritional intake. The antenatal period with the opportunities for regular contact with health professionals appears to be the ideal time and setting to institute the intervention which could maximize pregnant women's outcome and that of their baby by motivating them to make nutritional changes. The overall objective of the research was to assess the effect of nutrition education on the appropriate nutritional knowledge and practice of pregnant women.

DETAILED DESCRIPTION:
Adequate and balanced nutrition during gestation has been recognized as a prerequisite for a healthy pregnancy and birth outcomes and this is significantly determined by their nutritional knowledge and practice. This facility based single group pre-post quasi experimental study design was conducted with the objective of assessing the effect of nutrition education on the appropriate nutritional knowledge and practice of pregnant women. The study was conducted in five health facilities providing ANC (Antenatal Care) service in Asmara on 226 pregnant women. A predesigned and pretested questionnaire was used to collect data regarding nutritional knowledge via interview by trained data collectors during the pretest, immediate posttest and six weeks later. This study showed that the current intervention generally was effective in accomplishing improved knowledge and practice level of pregnant women. The simple nutrition education messages given to pregnant women using holistic approach of targeting all the major determinants in a sustained manner played a huge role in increasing their knowledge regarding nutrition during pregnancy. Knowledge regarding duration of iron supplementation was very low in this study. At the same time minor knowledge gap was seen in the sources of main food groups among pregnant women. The provided nutrition education also helped the pregnant women to improve dietary intake during pregnancy, although their adherence to iron supplements was decreased. Skipping meals and avoiding certain food items was also evident in this study. A reassuring concept is that food taboos and cultural factors were never the reasons that prevented women from consuming the food items. The educational intervention has shown more positive impact on increasing the scores regarding knowledge of appropriate nutrition during pregnancy for primigravida mothers than for multigravida mothers while the improvement in the dietary practice had no interaction with their socio-demographic characteristics. To sum up, attenuation of maternal and infant malnutrition may not be remote if pregnant women are well educated and counseled about nutrition during pregnancy. The study was conducted under limitations of not being able to control the possible effect of other sources like Television, books, magazines and radio broadcasting on the change in the knowledge and practice of pregnant women towards nutrition could not be controlled. Face to face interview may lead to social desirability bias which may in turn bring higher proportion of correct practice among pregnant women on the follow-up questioning (as the practice is self-reported).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who were on their first and second trimester of pregnancy and willing to participate in the study were included

Exclusion Criteria:

* Pregnant women who were sick at the time of the study and those who cannot communicate verbally.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 226 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2018-09-22 (Actual); Study Completion 2018-09-24 (Actual)

PRIMARY OUTCOMES:
knowledge level of pregnant women on nutrition and their appropriate nutrition-related practice after intervention | 6 weeks
  The two outcome variables in this study were the knowledge level of pregnant women and their appropriate nutrition-related practice after intervention. At the Data set of pregnant women the categorical data from the knowledge part of the data collection was recorded to dichotomous data of 1 and 0, where 1 is having the correct answer and 0 is for incorrectly answering. Practice components of the questionnaire of pregnant women were dichotomized to 1 and 0 as well, where 1 is having good practice and 0 is having no practice. Composite scores of knowledge and practice of each pregnant woman was computed. Mean scores of the knowledge (at pre, immediate post and 6 weeks later) and practice (at pre and 6 weeks later) of pregnant women were then calculated. The pregnancy specific NEC was the independent variable in this study. Co-variables on ANC clients were the demographics characteristics addition to source of information and frequency of ANC visits.

CONTACTS AND LOCATIONS:
Overall Officials: Lidia G Teweldemedhin, MSc, Principal Investigator — Lecturer
Locations (1):
- OCMHS, Asmara, Maekel Region, Eritrea

IPD SHARING:
Plan to Share IPD: No
I do not have plans to share my IPD

REFERENCES:
- [Background] Daba G, Beyene F, Fekadu H, Garoma W: Assessment of knowledge of pregnant mothers on maternal nutrition and associated factors in Guto Gida Woreda, East Wollega Zone, Ethiopia. Journal of Nutrition & Food Sciences 2013, 3(6):1.